CLINICAL TRIAL: NCT03227081
Title: Behavioral Modulation of Memory Traces: Influence of Sleep on Emotional Regulation and the Consolidation of Intrusive Memories
Brief Title: Behavioral Modulation of Intrusive Memories
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Dimitris Repantis, Dr. med., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SK 062016_rev
Record Dates: First submitted 2017-07-20; First posted 2017-07-24 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Intrusive Memories

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep (No Intervention): Sleep
- Sleep Deprivation (Experimental): Sleep Deprivation
  Interventions: Behavioral: Sleep Deprivation

INTERVENTIONS:
Behavioral: Sleep Deprivation — Sleep Deprivation
  Arms: Sleep Deprivation

SUMMARY:
The purpose of the study is to examine whether sleep affects the development of intrusive memories.

ELIGIBILITY:
Inclusion Criteria:

* healthy participants
* German on a native level

Exclusion Criteria:

* former or present psychiatric disorders
* physical illnesses
* history of trauma
* pregnancy or lactation period

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 101 (Actual)
Dates: Start 2017-07-17 (Actual); Primary Completion 2020-02-04 (Actual); Study Completion 2020-02-04 (Actual)

PRIMARY OUTCOMES:
Intrusive memories | seven consecutive days
  Intrusive memories measured with an intrusion diary

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Dimitris Repantis, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No